CLINICAL TRIAL: NCT00226759
Title: Double-Blind, Multicenter Phase 3 Study Comparing the Efficacy and Safety of OMS103HP With Vehicle in Patients Undergoing Allograft ACL Reconstruction
Brief Title: Efficacy and Safety of OMS103HP in Patients Undergoing Allograft Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C03511
Record Dates: First submitted 2005-09-26; First posted 2005-09-27 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Knee Injuries
Keywords: Anterior cruciate ligament reconstruction; ACL reconstruction
MeSH Terms: conditions — Knee Injuries | interventions — OMS 103HP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMS103HP irrigation solution (Experimental): Drug
  Interventions: Drug: OMS103HP
- vehicle irrigation solution (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS103HP — Maximum of 39 liters of OMS103HP irrigation solution over a maximum of 2 hours.
  Arms: OMS103HP irrigation solution
Drug: Vehicle — Maximum of 39 liters of vehicle irrigation solution over a maximum of 2 hours
  Arms: vehicle irrigation solution

SUMMARY:
The anterior cruciate ligament (ACL) is an important stabilizer of the knee. Orthopedic surgeons replace the torn ligament during ACL reconstruction surgery. Surgical trauma initiates an acute inflammatory response, including swelling and pain, that leads to restricted joint motion and loss of function. OMS103HP was designed to deliver targeted therapeutic agents directly to the surgical site during the arthroscopic procedure to inhibit inflammation and pain before they can begin.

The purpose of this study is to assess the effectiveness and safety of OMS103HP in improving knee function following ACL reconstruction. Secondary benefits being evaluated include reduced postoperative pain, improvement in knee range of motion and earlier return to work.

ELIGIBILITY:
Inclusion Criteria:

* 15 - 65 years of age
* In good general health with an ACL tear that occurred from 2 weeks to 18 months prior to the day of arthroscopic surgery
* Undergoing primary unilateral ACL reconstruction using an allograft (patellar tendon bone, Achilles tendon, tibialis tendon, or hamstring)
* Able to participate in the study rehabilitation protocol
* and other inclusion criteria

Exclusion Criteria:

* No allergies to any of the individual ingredients in OMS103HP
* No medications with the same activities as that of the active ingredients in OMS103HP for defined time intervals prior to and after surgery
* No associated knee injuries likely to interfere with evaluation of the study drug
* and other exclusion criteria

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2004-11; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Improvement in knee function | 30 days

SECONDARY OUTCOMES:
Decreased pain | 30 days
Improved range of motion | 30 days
Earlier return to work | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Houston, Study Director — Omeros Corporation
Locations (20):
- United States (18):
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Sports, Orthopedic and Rehabilitation Medicine Associates (S.O.A.R.), Redwood City, California
  - Stanford University, Stanford, California
  - Colorado Orthopedic Consultants, PC, Englewood, Colorado
  - American Clinical Research Services, Steamboat Springs, Colorado
  - University of Florida, Gainesville, Florida
  - Southeastern Center for Clinical Trials, Atlanta, Georgia
  - Minnesota Sports Medicine, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio
  - University Orthopedics Center, Altoona, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Texas Orthopedics, Austin, Texas
  - Round Rock Orthopedics, Round Rock, Texas
  - Unlimited Research, San Antonio, Texas
  - Hill Country Sports Medicine, San Marcos, Texas
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
- Canada (2):
  - Rouge Valley Health Systems, Ajax, Ontario
  - Hotel Dieu Grace Hospital, Windsor, Ontario